CLINICAL TRIAL: NCT03033316
Title: A Phase I-IIa, Open Label, Multi-Center, Dose Escalating Study to Evaluate the Safety of Intravenous Pegylated Liposomal Dexamethasone Sodium Phosphate (Oncocort) as Monotherapy in Patients With Previously Treated Progressive Multiple Myeloma
Brief Title: A Evaluation of the Safety of Oncocort IV Pegylated Liposomal Dexamethasone Phosphate in Patients With Progressive Multiple Myeloma
Acronym: AMETHYST
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Patient enrolment issues
Sponsor: Enceladus Pharmaceuticals BV (Industry)
Collaborators: University Hospital, Aachen (Other); Accelovance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-097
Record Dates: First submitted 2017-01-03; First posted 2017-01-26 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Liposomal Dexamethasone; Targeted Drug Delivery
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IV Liposomal Dexamethasone (Experimental): IV Liposomal Dexamethasone given 1 to 4 times in total over period of maximally 4 weeks
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone

SUMMARY:
Oncocort Dexamethasone sodium phosphate encapsulated in so-called 'long-circulating' PEGylated liposomes is in development with the prospect of providing enhanced and prolonged lesion uptake of dexamethasone and therefore increased therapeutic benefit over existing formulations of dexamethasone in Multiple Myeloma. The current trial is a first-in-man study with Oncocort monotherapy with the objective to assess safety, tolerability, efficacy and dose response after short-term treatment with repeated infusions.

DETAILED DESCRIPTION:
This open label multicenter study will evaluate the safety and efficacy of I.V. Oncocort Dexamethasone sodium phosphate given as a short term induction therapy in Multiple Myeloma patients. It consist of a Phase 1 part with a maximum number of 5 ascending dose levels while additional patients will be treated in the Phase 2a part with the recommended phase 2 dose to obtain additional safety data and preliminary efficacy data in multiple myeloma patients. For the dose escalation phase 1 part, 3 patients per dose level will be enrolled. If one patient reaches DLT, another 3 patients will be enrolled in the same dose level. If two or more patients reach DLT in one dose level, maximum tolerated dose (MTD) is defined at the last dose level beneath DLT. Not more than 5 dose level groups are anticipated for this part of the study. MTD will be the Recommended Phase II Dose (RPTD) for the phase IIa part of the study. For the phase 2a part, 7 additional patients will be enrolled at the RPTD dose level, bringing the total number of patients monitored for responses at this dose level to at least 10.

ELIGIBILITY:
Inclusion Criteria

1. Previously diagnosed symptomatic MM according to International Myeloma Working Group (IMWG) criteria 1.1. Previously treated with at least two therapy lines including at least one proteasome-inhibitor and at least one immunomodulatory drug 1.2. Relapse after or progressive disease under last therapy according to IMWG criteria.
2. At least 18 years old
3. Measurable disease (M-protein and/or free light chains) in serum and/or urine
4. Willing and able to comply the study protocol visits and assessments
5. Willing to use highly effective methods of birth control (see section 7.1.3)
6. Written informed consent prior to study participation

Exclusion Criteria:

1. Types of Multiple Myeloma previously shown to be irresponsive to dexamethasone monotherapy during the last 6 months
2. Plasma cell leukemia
3. Subject with positive hepatitis panel (including hepatitis B surface antigen [HBsAg], and / or anti-hepatitis B core antibodies, and / or hepatitis C virus antibody [anti-HCV]), and / or a positive HIV antibody screen
4. Severe abnormal organ function function or laboratory results at the time of the Screening Visit: WBC <3.0 g/L, ANC <1.5 G/L, PLT <50 G/L, Sodium <135 mmol/L or >150 mmol/L, potassium <3.5 mmol/L or >5.5 mmol/L, calcium <2.0 mmol/L or > 2.9mmol/L, phosphorus <0.8 mmol/L, total bilirubin >1.5x ULN, AP >2.5x ULN, gammaGT >3x ULN, ALT >3x ULN, CK >2.5x ULN, Creatinine >2x ULN, fasting glucose >250 mg/dL, albumin <3 g/dL, cholesterol > 300 mg/dL
5. Treatment with oral or injectable (including intra-articular) corticosteroids (CS) within 4 weeks prior to Screening Visit. Inhaled and dermal corticosteroid formulations are allowed
6. Subjects who have received a chemotherapeutic treatment cycle including dexamethasone within 4 weeks prior to the Screening Visit
7. Known sensitivity to any component of the study drug or previous hypersensitivity reaction or other clinically significant reaction to intravenous medications, biologic therapy or IV radiocontrast agents
8. Active infection requiring systemic treatment
9. Planned major surgery during the study period or had undergone major surgery within 30 days prior to the Screening visit
10. Pregnancy or breastfeeding
11. Any clinically significant hepatic, renal, cardiac, pulmonary, gastrointestinal, metabolic or endocrine disturbances, other medical or psychiatric condition, or clinically relevant abnormal values on any investigation, in the opinion of the Investigator, that could make the subject unsuitable for the study, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study, including severe neuropathies or other painful conditions that might interfere with pain evaluation
12. Participation in another clinical investigation less than 4 weeks prior to inclusion
13. The subject has a history of any other illness, which, in the opinion of the Investigator, might pose an unacceptable risk by administering study medication.
14. The subject has any current or past medical condition and/or required medication to treat a condition that could affect the evaluation of the study
15. The subject is unwilling or unable to follow the procedures outlined in the protocol
16. The subject is mentally or legally incapacitated
17. Persons who are in a relationship of dependence to the Investigator or the Sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Week 8

SECONDARY OUTCOMES:
Response according to IMWG Criteria | 4 and 8 weeks after 1st dose
Percentage change of myeloma-related measures | up to 8 weeks after 1st dose
Quality of life questionnaire | up to 8 weeks after 1st dose
Peak Plasma Concentration (Cmax) | during 1st 4 weeks
Area under the plasma concentration versus time curve (AUC) | during 1st 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Wilop, MD, Principal Investigator — RWTH University Clinic Aachen

IPD SHARING:
Plan to Share IPD: No